CLINICAL TRIAL: NCT01219140
Title: A Randomized, Placebo-Controlled, Double-Blind, Parallel Design Trial to Evaluate the Safety and Efficacy of Pomegranate Extract Capsules in Post-Menopausal Subjects With Decreased Bone Mineral Density
Brief Title: Pomegranate Extract Biomarker Study in Osteopenic Women
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: POM Wonderful LLC (Industry)
Responsible Party: POM Wonderful LLC
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: POM 2010-001
Record Dates: First submitted 2010-10-08; First posted 2010-10-13 (Estimated); Last update posted 2010-10-13 (Estimated); Status verified 2010-10

CONDITIONS: Osteopenic Women
Keywords: POMx; Osteopenia; postmenopausal women; Pomegranate
MeSH Terms: conditions — Bone Diseases, Metabolic

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- 2 POMx Capsules (Experimental): 2 POMx Capsules daily
  Interventions: Dietary Supplement: 2 POMx Capsules
- 2 placebo Capsules (Placebo Comparator): 2 placebo Capsules daily
  Interventions: Dietary Supplement: 2 placebo Capsules

INTERVENTIONS:
Dietary Supplement: 2 POMx Capsules — 2 POMx Capsules daily
  Arms: 2 POMx Capsules
Dietary Supplement: 2 placebo Capsules — 2 placebo Capsules daily
  Arms: 2 placebo Capsules

SUMMARY:
Treatment of post-menopausal subjects (with decreased bone mineral density) with pomegranate extract capsules will produce statistically significant changes in biomarkers for bone resorption and formation when compared to subjects receiving placebo.

ELIGIBILITY:
Inclusion Criteria:

* Postmenopausal women (having had their last menstrual period within the past 15 years and an appropriate serum FSH value) 45-65 years of age;
* The subject must have a T score of -1 to -2.5 at the lumbar spine or proximal femur;
* All clinical safety laboratory values at screening and randomization must be either within the reference range or be determined by the investigator and the sponsor to be abnormal, but not clinically significant;
* The patient must have provided written informed consent.

Exclusion Criteria:

* The subject has any of the following conditions: connective tissue disease, history of clinically significant renal, hepatic pulmonary, cardiovascular, cerebrovascular, gastrointestinal, metabolic, hematological, endocrinological, urological, immunological, neurologic or psychiatric disorders, unless approved by the sponsor on a case by case basis;
* The subject has a positive test result for Hepatitis B surface antigen or antibody to hepatitis C virus at Screening;
* The subject has a known history of infection with the human immunodeficiency virus (HIV); -
* The subject has used bisphosphonate or fluoride therapy within the past 12 or 24 months, respectively;
* The subject has used denosumab within the past 24 months;
* The subject has used tibolone, parathyroid hormone (or any of its derivatives), systemic glucocorticoids or inhaled glucocorticoids, anabolic steroids or testosterone within the past 6 months;
* The subject has used estrogens, selective estrogen receptor modulators, calcitonin or calcitriol within the past 3 months;
* The subject has hyperparathyroidism, hypoparathyroidsim, hyperthyroidism, hypothyroidism, hypocalcemia, rheumatoid arthritis, paget's disease of bone, osteomalacia;
* The subject has had a bone fracture within the past year;
* The subject has acute or chronic disease requiring frequent changes in medications or dosages of chronic therapy;
* A history of alcoholism within the last 2 years or a current history of imbibing 3 or more units of alcohol per day. (1 unit is equivalent to 1 glass of wine, 1 pint of beer, or 1 shot of hard liquor);
* The subject has participated in another study with an investigational drug or device during the 30 days prior to study entry;
* The subject has a condition interfering with his ability to provide informed consent or comply with study instructions, or the patient has a condition, which might confound the interpretation of the study result;
* The subject has a condition endangering herself if she were to participate in this trial

Ages: 45 Years to 65 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 64 (Actual)
Dates: Start 2010-05; Primary Completion 2010-10 (Actual); Study Completion 2010-10 (Actual)

PRIMARY OUTCOMES:
Biomarkers | Throughout study
  To evaluate the impact of pomegranate extract capsules on urinary N-terminal telopeptide (NTX) and serum procollagen type 1 amino-terminal propeptide (P1NP), in post-menopausal women with decreased bone mineral density

SECONDARY OUTCOMES:
Number of Participants with Adverse Events as a Measure of Safety and Tolerability | Throughout study
  Incidence of adverse events Changes in vital signs or laboratory values

CONTACTS AND LOCATIONS:
Locations (1):
- SeaView Research, Inc., Miami, Florida, United States